CLINICAL TRIAL: NCT02695277
Title: Combined Endoscopic Epicardial and Percutaneous Endocardial Ablation Versus Repeated Catheter Ablation in Persistent and Longstanding Persistent Atrial Fibrillation
Acronym: CEASE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Collaborators: Cardialysis BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP2015-1
Record Dates: First submitted 2015-12-14; First posted 2016-03-01 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation; Persistent and Longstanding Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Persistent and Longstanding Persistent AF; Hybrid Procedure; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hybrid Procedure (Experimental): Endoscopic epicardial surgical ablation (first stage) combined with endocardial catheter ablation (second stage) performed between 91 and 180 days post index procedure.
  Interventions: Device: AtriCure Bipolar System; Device: AtriClip® PRO LAA Exclusion System; Device: Endocardial Ablation with Catheter
- Catheter Procedure (Active Comparator): Standard catheter ablation with pulmonary vein (PV) isolation (minimum lesion set) and optional additional lesions (index procedure). When required due to AF recurrence, ablation may be repeated within 6 months after the index-procedure according to clinical indications and consistent with the Heart Rhythm Society (HRS)/European Heart Rhythm Association (EHRA)/European Cardiac Arrhythmia Society (ECAS) Consensus Statement
  Interventions: Device: Standard Endocardial Ablation with Catheter; Device: Repeated Endocardial ablation(s)

INTERVENTIONS:
Device: AtriCure Bipolar System
  Arms: Hybrid Procedure
Device: Standard Endocardial Ablation with Catheter
  Arms: Catheter Procedure
Device: AtriClip® PRO LAA Exclusion System
  Arms: Hybrid Procedure
Device: Endocardial Ablation with Catheter
  Arms: Hybrid Procedure
Device: Repeated Endocardial ablation(s)
  Arms: Catheter Procedure

SUMMARY:
This is a prospective, randomized (2:1) multicenter trial to investigate the optimal treatment of Persistent and Longstanding Persistent AF referred for Radiofrequency (RF) ablation.The study objective is to compare the efficacy and safety of two interventional approaches, in preventing the recurrence of AF in symptomatic, drug refractory patients with persistent or longstanding persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a history of symptomatic Persistent AF and a left atrium (LA) > 4cm or Long Standing Persistent AF as defined by the HRS/EHRA/ECAS expert consensus statement
2. Patient is refractory to or intolerant of at least one antiarrhythmic drug (class I or III)
3. Patient is mentally able and willing to give informed consent

Exclusion Criteria:

1. Patient has longstanding persistent AF > 10 years
2. Patient presenting with paroxysmal AF
3. Patient with persistent AF and a LA-diameter ≤ 4cm
4. AF is secondary to electrolyte imbalance, thyroid disease, or other reversible or non-cardiovascular cause
5. Patient underwent previous ablation procedure or heart surgery
6. Patient needs other cardiac surgery procedures besides AF treatment (valve, coronary, others)
7. Contraindication for either catheter ablation or epicardial surgery (including, but not limited to: previous thoracic radiation, previous perimyocarditis, Previous cardiac tamponade, Pleural adhesions, Prior thoracotomy)
8. Body mass index > 35
9. LA Diameter > 6 cm
10. Left ventricular ejection fraction < 30 %
11. Severe mitral regurgitation (>II)
12. Patient unable to undergo TransEsophageal Echocardiogram (TEE)
13. Presence of LA thrombus by TEE, CT scan, MRI or angiography
14. History of cerebrovascular disease, including stroke or transient ischemic attack (TIA) within 6 months prior to enrollment
15. Active infection or sepsis
16. Other clinical conditions precluding inclusion (e.g., organ disease, disturbances of hemostasis)
17. Contraindication to anticoagulant therapy, or inability to comply with anticoagulant therapy
18. Pregnancy, planned pregnancy or breastfeeding
19. Life expectancy is less than 12 months
20. Patient is involved in another study involving an investigational drug or device

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects free from documented Atrial Fibrillation (AF), Atrial Flutter (AFL) or Atrial Tachycardia (AT) episodes > 30 seconds in duration through 12 months follow-up, in the absence of Class I or III Antiarrhythmic Drugs (AADs). | Through 12-months post the Endocardial procedure (Hybrid Procedure) or last allowed Catheter Ablation(Catheter Procedure)

SECONDARY OUTCOMES:
Number of subjects free from documented AF, AFL or AT episodes > 30 seconds in duration through 24 and 36 months follow-up, in the absence of Class I or III AADs. | Through 24- and 36-months post the Endocardial procedure (Hybrid Procedure) or last allowed Catheter Ablation(Catheter Procedure)

OTHER OUTCOMES:
Composite major complications | Up to 180 days (6-months) post index procedure

CONTACTS AND LOCATIONS:
Locations (12):
- Czechia (2):
  - Dr Tomáš Ostřížek, Brno
  - Czech Budejovice Hospital, Inc., České Budějovice
- Germany (7):
  - Cardiovascular Center Bad Neustadt, Bad Neustadt an der Saale
  - Schüchtermann-Schiller'sche Kliniken Herzzentrum Osnabrück, Bad Rothenfelde
  - Heart Center Leipzig, Leipzig
  - Klinikum Ludwigsburg, Ludwigsburg
  - Peter Osypka Heart Center Munich, Munich
  - Kliniken Sindelfingen, Sindelfingen
  - Sana Heart Center Stuttgart, Stuttgart
- St. Antonius Hospital, Nieuwegein, Netherlands
- Central Clinical Hospital of the Ministry of Interior, Warsaw, Poland
- Northern General Hospital, Sheffield, United Kingdom

REFERENCES:
- [Derived] Doll N, Weimar T, Kosior DA, Bulava A, Mokracek A, Monnig G, Sahu J, Hunter S, Wijffels M, van Putte B, Rub N, Nemec P, Ostrizek T, Fransen E, Suwalski P. Durable effectiveness and safety of hybrid ablation versus catheter ablation: 2-year results from the randomized CEASE-AF trialdagger. Eur J Cardiothorac Surg. 2025 Jul 1;67(7):ezaf146. doi: 10.1093/ejcts/ezaf146. PMID 40711852